CLINICAL TRIAL: NCT06451562
Title: A Controlled Study to Compare the Effect of Regional Anesthesia by an Erector Spine Plane Block and Intravenous Infusion of Lidocaine on the Rate of Intravenous Morphine Use After Scoliosis Repair Surgery
Brief Title: Effect of Regional Anesthesia or Intravenous Infusion of Lidocaine on Morphine Use After Scoliosis Repair Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Zoya Haitov Ben Zikri, Manager of the anesthesia unit, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0008-24-ASF
Record Dates: First submitted 2024-05-21; First posted 2024-06-11 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): This group will serve as a control - the patients will receive general anesthesia according to the standard protocol for general anesthesia in this study. Upon the end of the surgery, patients will begin receiving analgesics and anti-nausea treatment according to the standard protocol in this study.
- Erector spinae plane block (Active Comparator): Patients will receive general anesthesia according to the standard protocol for general anesthesia in this study. After induction for anesthesia, before the start of the surgery, the anesthesiologist will perform an ultrasound guided ESP block, according to the ultrasound guided erector spinae plane block protocol
  Interventions: Drug: Lidocaine
- Lidocaine (Active Comparator): Patients will receive general anesthesia according to the standard general anesthesia protocol for this study. In addition, after induction of anesthesia, patients will begin receiving an intravenous infusion of lidocaine at a dose of 0.5 mg per kg per hour, and will continue to receive the infusion after surgery for a total of 24 hours.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — a local anesthetic drug of the amino amide type
  Other Names: Lignocaine; Xylocaine
  Arms: Erector spinae plane block; Lidocaine

SUMMARY:
The goal of the surgical correction of scoliosis is to prevent progression of the curve or progression of restrictive lung disease. After scoliosis surgery, patients experience severe pain. The standard treatment for pain relief after scoliosis surgery is the administration of opiates. However, treatment with these substances involves side effects such as respiratory depression, nausea and vomiting, inhibition of bowel activity and itching. To lower the dose of opiates, different types of painkillers and other techniques can be added.

The purpose of the study is to compare the effect of instillation of lidocaine (which is an analgesic and anti-inflammatory) or regional anesthesia using Erector spinae plane on the dose of morphine consumption, the intensity of pain, the side effects and the quality of recovery during the first 48 hours after surgery to repair scoliosis.

DETAILED DESCRIPTION:
The goal of the surgical correction of scoliosis is to prevent progression of the curve or progression of restrictive lung disease. After scoliosis surgery, patients experience severe pain. The standard treatment for pain relief after scoliosis surgery is the administration of opiates. The opiate that is usually used after scoliosis repair surgery to correct scoliosis is morphine. It is given independently by the patients using the patient-controlled analgesia device. However, treatment with these substances involves side effects such as respiratory depression, nausea and vomiting, inhibition of bowel activity and itching. To lower the dose of opiates, different types of painkillers and other techniques can be added.

The purpose of the study is to compare the effect of instillation of lidocaine (which is an analgesic and anti-inflammatory) or regional anesthesia using Erector spinae plane on the dose of morphine consumption, the intensity of pain, the side effects and the quality of recovery during the first 48 hours after surgery to repair scoliosis.

Patients will be randomized to one of 3 groups. The patients do not know which group they belong to.

Group C - control - the patients will receive general anesthesia according to the standard protocol for general anesthesia in this study.

Group B - ESP block - patients will receive general anesthesia according to the standard protocol for general anesthesia in this study. And then the anesthesiologist will perform an ultrasound-guided ESP block

Group L - Lidocaine - Patients will receive general anesthesia according to the standard protocol for general anesthesia for this study. In addition, after induction of anesthesia, patients will begin receiving an intravenous infusion of lidocaine and will continue to receive the infusion after surgery for a total of 24 hours.

The patients will be connected to the PCA device by the anesthetists before leaving for recovery unit. The patients will receive an explanation before and after the operation to press the PCA bolus only if there is strong bursting pain. 48 hours after the surgery, the PCA will be stopped and patients will receive other pain relievers as needed.

Patient report data on the level of pain and nausea will be collected 1, 6, 12, 24, and 48 hours after the end of the surgery. Data will also be collected on the maximum dose of morphine that the patient received from the PCA pump 24 and 48 hours after the end of the operation, the time of the first bowel movement and the time of the first walk, as well as demographic data of the patients. The QOR-15 questionnaire to check the quality of recovery will be filled out by the patients 72 hours after the end of the surgery

ELIGIBILITY:
Inclusion Criteria:

Patients over the age of 12 with normal cognition, who are scheduled to undergo surgery to correct scoliosis and treatment with IV PCA independently for pain relief after surgery; The patients' parents/guardian (in the case of a minor) or the patient himself (in the case of an adult) signed an informed consent form for participation in the study; Patients should be able to operate the PCA device independently

Exclusion Criteria:

Patients who do not agree to participate in the study even if their parents signed an informed consent

Patients who are unable to operate the PCA device independently

Patients under treatment with opioids or cannabis for chronic pain for more than a month;

Drug use of any kind;

Alcoholism;

Patients with depression, anxiety or post-trauma;

Moderate-severe insufficiency of one of the systems - respiratory/cardiac/hepatic/renal;

Sensitivity to one of the drugs in the research protocol.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | 48 hours after surgery
  Dosage of morphine consumption in milligrams that the patients will consume in by pressing on the PCA device in the first 48 hours after surgery to correct scoliosis

SECONDARY OUTCOMES:
Quality of recovery | 72 hours after surgery
  The patient will fill the QOR15 questionnaire for Quality of recovery
Pain intensity, | 48 hours after surgery. The pain will be monitored at 1, 6, 12, 24 and 48 hours after the surgery.
  Monitoring the effect of treatments on pain intensity during the first 48 hours after surgery. Using patients' reported NRS scale 0-10 with 0 meaning no pain at all and 10 meaning the worst imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bar Yehuda, PhD, Study Director — Shamir (Asaf Harofe) medical center
Locations (1):
- Shamir (Asaf Harofe) Medical Center, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: No